CLINICAL TRIAL: NCT05738694
Title: A Multicenter Randomized Controlled Clinical Study of Neoadjuvant Combination of Axitinib Plus PD-1 Monoclonal Antibody to Improve Disease Free Survival of Patients With Renal Cell Carcinoma
Brief Title: Neoadjuvant of Axitinib Plus PD-1 to Improve Disease Free Survival of Patients With Renal Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ZHOU FANGJIAN (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, ZHOU FANGJIAN, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-FXY-518
Record Dates: First submitted 2023-01-11; First posted 2023-02-22 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Renal Cell Carcinoma; Neoadjuvant
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Axitinib; toripalimab; Nephrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neoadjuvant group (Experimental): Neoadjuvant group will be given the neoadjuvant combination of axitinib plus Toripalimab + nephrectomy
  Interventions: Drug: Axitinib plus Toripalimab; Procedure: nephrectomy
- Control group (Active Comparator): The control group will be given nephrectomy alone.
  Interventions: Procedure: nephrectomy

INTERVENTIONS:
Drug: Axitinib plus Toripalimab — Preoperative treatment with axitinib will be given for 3 months, 5 mg twice daily, orally. Preoperative treatment with Toripalimab will be given for 4 cycles (3 weeks considered one cycle), 240 mg, Q3W.
  Other Names: nephrectomy
  Arms: Neoadjuvant group
Procedure: nephrectomy — nephrectomy

SUMMARY:
The study included 298 RCC patients who were at high risk for recurrence after nephrectomy (T2G3-4 or T3-4 or N1). They were randomly divided to receive axitinib plus PD-1 + surgery or surgery alone at a ratio of 1:1, so as to determine the efficacy of the neoadjuvant combination of axitinib plus PD-1.

DETAILED DESCRIPTION:
Given the good results of TKI plus PD-1 in our previous cases and its good effect on advanced RCC, we plan to eliminate tumor micrometastases and improve anti-tumor immunity with the neoadjuvant combination of axitinib plus PD-1, so as to improve patient outcomes. The study included 298 RCC patients who were at high risk for recurrence after nephrectomy (T2G3-4 or T3-4 or N1). They were randomly divided to receive axitinib plus PD-1 + surgery or surgery alone at a ratio of 1:1, so as to determine the efficacy of the neoadjuvant combination of axitinib plus PD-1 and provide evidence-based medical evidence for clinical perioperative treatment of these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily agree to participate in this study and sign the informed consent form;
2. Males or females between 18 years old and 80 years old;
3. Diagnosed as clear cell carcinoma or renal cell carcinoma predominantly composed of clear cell carcinoma through histopathological examination
4. CT or MRI clinical staging is T2G4 or T2 with sarcomatoid differentiation, T3-4, N1;
5. ECOG performance status: 0 or 1 point;
6. Sufficient heart, bone marrow, liver, and kidney functions:

Cardiac function: Cardiac function class 0-2; Blood routine test: WBC≥3.5×10^9/L, absolute neutrophil count ≥1.5×10^9/L, PLT≥75.0×10^9/L, HGB≥80g/L; Liver function: Total bilirubin ≤1.5×upper limit of normal (ULN), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5×ULN; Renal function: GFR ≥ 45 ml/min.

Exclusion Criteria:

1. With distant metastasis
2. Severe liver and renal dysfunction, combined with other serious diseases;
3. Serious cardiovascular disease, including any of the following: myocardial infarction or arteritis or venous thrombosis (such as pulmonary embolism) in the past 1 year;
4. Severe/unstable angina pectoris; uncontrolled hypertension;
5. Class III or IV heart failure by New York Heart Association (NYHA) Functional Classification;
6. Ventricular arrhythmia requiring drug treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Estimated)
Dates: Start 2023-04-19 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
disease-free survival (DFS) | 2 years
  To evaluate the efficacy of the neoadjuvant combination of axitinib plus PD-1 in improving the 2-year disease-free survival (DFS) in RCC patients with high-risk for recurrent (T2G3-4 or T3-4, or N1). Disease-free survival (DFS) is defined as time from registration to disease progression or death.

SECONDARY OUTCOMES:
The cancer-specific survival (CSS) | 3 years
  cancer specific survival (CSS) is defined as the period between the date of randomization and the date of death from renal cancer.
overall survival (OS) | 3 years
  overall survival (OS) is defined as the period between the date of randomization and the date of death from any cause
objective response rate (ORR) | 3 years
  CR and PR rate as assessed by RECIST 1.1
major pathological response (MPR) | 3 years
  MPR (≤10% viable malignant cells per local pathology assessment)
adverse event management | 3 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Fangjian Zhou, Professor, Principal Investigator — Director of Dept. of Urology, Sun Yat-sen University Cancer Center
Locations (8):
- China (8):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - Peking University First Hospital, Beijing
  - Sun Yat-sen University Cancer Center, Guangzhou
  - Anhui Provincial Hospital, Hefei
  - Fudan University Cancer Hospital, Shanghai
  - West China Hospital, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin
  - The First Affiliated Hospital of Zhengzhou Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: No